CLINICAL TRIAL: NCT04159051
Title: Phase II Studie Zur Hyperthermen Salvage-Radiotherapie Bei Prostatakarzinompatienten Mit Biochemischem Rezidiv Nach Prostatektomie
Brief Title: Charité HT-Prostate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Pirus Ghadjar, Head of Hyperthermia Unit, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA2/110/15
Record Dates: First submitted 2019-11-06; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer; Recurrence
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined regional hyperthermia and salvage radiotherapy (Experimental)
  Interventions: Device: Regional Hyperthermia

INTERVENTIONS:
Device: Regional Hyperthermia — Regional hyperthermia 1-2×/week to a total number of 7-10 treatments combined with salvage radiotherapy to a total dose of 70 Gy over 7 weeks

SUMMARY:
The combination of regional hyperthermia and salvage radiotherapy is being tested in patients with biochemically recurrent prostate cancer after radical prostatectomy.

DETAILED DESCRIPTION:
Current studies on salvage radiotherapy (sRT) for biochemically recurrent prostate cancer after radical prostatectomy investigate timing, dose-escalation and androgen deprivation therapy (ADT) for recurrent prostate cancer. These approaches could either be limited by radiation-related susceptibility of the anastomosis or by suspected side-effects of ADT. A phase II protocol was developed to investigate the benefit and tolerability of regional hyperthermia with moderately dose-escalated sRT. The study hypothesis is that hyperthermic sRT is a safe and feasible salvage treatment modality. The primary endpoint is safety measured by frequency of grade 3+ genitourinary (GU) and gastrointestinal (GI) adverse events (AE) according to Common Toxicity Criteria (CTC) version 4. Feasibility is defined by number of hyperthermia treatments (n ≥ 7) and feasibility of sRT according to protocol. Target volume delineation is performed according to the EORTC guidelines. sRT is administered with single doses of 2 Gy 5×/week to a total dose of 70 Gy to the prostate bed, or alternatively the total dose only to the area of highest risk and a lower dose to the remaining prostate bed using a simultaneous boost (SIB) technique. Regional hyperthermia is given 2×/week to a total of 10 treatments. German centres participate in the phase II trial using intensity modulated RT (IMRT), volumetric modulated arc technique (VMAT) or tomotherapy. The initiating centres were participants of the SAKK 09/10 study, where the same patient criteria and target volume definition (mandatory successful performed dummy run) were applied insuring a high standardisation of the study procedures.

The introduced phase II study implements modern sRT and regional hyperthermia. If the phase II study is found to be safe and feasible, a multicenter phase III study might be performed to test whether the addition of regional hyperthermia to dose-intensified sRT improves biochemical control.

ELIGIBILITY:
Inclusion Criteria:

1. Lymph node negative adenocarcinoma of the prostate treated with radical prostatectomy at least 12 weeks before randomization. Tumour stage pT2a-3b, R0-1, pN0 or cN0 according to the UICC TNM 2009; Gleason score available.
2. PSA progression after prostatectomy defined as two consecutive rises with the final PSA > 0.1 ng/ml or three consecutive rises. The first value must be measured at least 4 weeks after radical prostatectomy.
3. PSA at randomization ≤ 2 ng/ml.
4. No evidence of macroscopic local recurrence or metastatic disease on pre-sRT-MRI (magnetic resonance imaging; with i.v. contrast) or pre-sRT-CT (multislice computed tomography with i.v. and oral contrast) of the abdomen and pelvis assessed within 16 weeks prior to randomization.
5. WHO performance status 0-1 at randomization.
6. Age at randomization between 18 and 80 years.
7. Informed consent.

Exclusion Criteria:

1. Persistent PSA value 4-20 weeks after radical prostatectomy > 0.4 ng/ml.
2. Palpable mass in the prostatic fossa, unless histology proves no evidence of recurrence.
3. Pelvic lymph node enlargement >1 cm in short axis diameter of the abdomen and pelvis (cN1), unless the enlarged lymph node is sampled and negative.
4. Presence or history of bone metastases. Bone scan is mandatory in cases of clinical suspicion (e.g., bone pain).
5. Other malignancies within five years before planned sRT; non-melanoma skin cancers are allowed.
6. ADT or bilateral orchiectomy.
7. Previous pelvic radiotherapy.
8. Hip prosthesis.
9. Metal clusters/markers and patients with a pacemaker.
10. Severe or active co-morbidities impairing the feasibility of hyperthermia or dose intensified sRT including (but not exclusively limited to):

    * chronic inflammatory bowel disease
    * acute bacterial or fungal infection requiring intravenous antibiotics at the time of randomization
    * unstable angina pectoris and/or congestive heart failure requiring hospitalization within the last 6 months
    * transmural myocardial infarction within the last 6 months
    * chronic obstructive pulmonary disease exacerbation or other respiratory disorders requiring hospitalization or precluding planned treatment within the study at the time of randomization
    * psychiatric disorder precluding understanding of information on trial-related topics, giving informed consent or filling out QoL questionnaires
11. Concurrent treatment with other experimental drugs or other anti-cancer therapy; treatment in a clinical trial within 30 days prior to trial entry.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Acute grade 3+ adverse events | up to three months after end of treatment
  Measured according to CTCAE version 4.

SECONDARY OUTCOMES:
Late adverse events | up to 36 months after end of treatment
  According to CTCAE version 4.
Quality of life (QoL) assessment | up to 36 months after end of treatment
  Using EORTC questionnaires
Biochemical progression-free survival | up to 36 months after end of treatment
  PSA-rise > 0.4 ng/ml or increasing PSA-level where the initial PSA-level is above 0.4 ng/ml.
Clinical progression-free survival | up to 36 months after end of treatment
  Occurrence of a local recurrence, regional recurrence or distant metastasis. Clinical progression-free survival is defined as the time between trial inclusion and occurrence of clinical progression, start of a new androgen deprivation therapy (see below) or death. Patients without event will be censored at the time of last follow-up.
Time without androgen deprivation therapy (ADT), i.e., time until initiation of ADT | up to 36 months after end of treatment
  The time from trial inclusion until start of a new androgen deprivation therapy. Patients without new ADT will be censored at the time of last follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Charité Universitätsmedizin Berlin, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muller AC, Zips D, Heinrich V, Lamprecht U, Voigt O, Burock S, Budach V, Wust P, Ghadjar P. Regional hyperthermia and moderately dose-escalated salvage radiotherapy for recurrent prostate cancer. Protocol of a phase II trial. Radiat Oncol. 2015 Jul 8;10:138. doi: 10.1186/s13014-015-0442-4. PMID 26152590